CLINICAL TRIAL: NCT02457000
Title: Sleep, Circadian Rhythm & Skin Health
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Kevin Cooper, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 12-14-23
Record Dates: First submitted 2015-03-18; First posted 2015-05-29 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Healthy; Psoriasis; Eczema; Acne
Keywords: Sleep; Skin; Circadian Rhythm
MeSH Terms: conditions — Psoriasis; Eczema; Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Skin, blood, urine, saliva and hair follicle samples may be collected from volunteers to look at various markers related to sleep, the circadian rhythm and skin disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal, healthy volunteers: Normal, healthy volunteers without any skin pathology will be asked to undergo various procedures to evaluate their sleep and skin health.
- Volunteers with skin pathology: Volunteers with skin pathology including but not limited to eczema, psoriasis, acne, and other inflammatory dermatoses will be asked to undergo various procedures to evaluate their sleep and skin health.

SUMMARY:
The purpose of this study is to explore the mechanisms behind how sleep quality may affect skin aging, skin integrity and skin disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 18 years and above
* Capable of giving informed consent
* Adults who are either healthy, normal volunteers or those with a skin disease including but not limited to eczema, psoriasis, acne or other inflammatory dermatoses
* Fitzpatrick Skin Type I-VI
* In good general health
* Willing to cooperate with study instructions

Exclusion Criteria:

* Volunteers 18 years or younger
* Any serious medical or physical condition that would cause the subject significant discomfort with study procedures
* Women who are pregnant, nursing, or who may become pregnant in the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults from Northeast Ohio who are either healthy, normal volunteers or have skin pathology including but not limited to eczema, psoriasis, acne, and other inflammatory dermatoses
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Analysis of Sleep Pattern via Actigraphy, Polysomnography & Questionnaires | 7-14 days
  The volunteers may be asked to wear a wrist actigraph to measure movement. This watch would be worn for 24 hours per day for 7-14 days. The volunteer may also be asked to fill out questionnaires regarding their sleep patterns. Note: Other methods of assessing sleep patterns may also be used including a portable polysomnogram or a standard, overnight sleep study.
Evaluation of skin (both in terms of skin aging and skin disease) | Only once during the study or at specific time points depending on what other procedures are being performed
  The volunteers may have their skin evaluated for skin aging using the SCINEXA tool. Volunteers with psoriasis may have their skin evaluated via PASI and/or PGA assessments. Volunteers may have photographs taken to compare clinical appearance with laboratory and research findings.

SECONDARY OUTCOMES:
Sample Analysis (from skin, blood, urine, saliva and hair follicle samples) | Only once during the study or at specific time points depending on what other procedures are being performed
  Skin, blood, urine, saliva and hair follicle samples may be collected from some volunteers to look at various markers related to sleep, the circadian rhythm and skin disease.
Skin Barrier Recovery (via TEWL measurement) | Only once during the study or at specific time points depending on what other procedures are being performed
  Skin barrier recovery via Transepidermal Water Loss (TEWL) measurement may be assessed in some volunteers.
MED Testing & Recovery from UV-induced erythema | 24 hours
  MED Testing & Recovery from UV-induced erythema may be assessed in some volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Oyetakin-White P, Suggs A, Koo B, Matsui MS, Yarosh D, Cooper KD, Baron ED. Does poor sleep quality affect skin ageing? Clin Exp Dermatol. 2015 Jan;40(1):17-22. doi: 10.1111/ced.12455. Epub 2014 Sep 30. PMID 25266053
- [Background] Rogiers V; EEMCO Group. EEMCO guidance for the assessment of transepidermal water loss in cosmetic sciences. Skin Pharmacol Appl Skin Physiol. 2001 Mar-Apr;14(2):117-28. doi: 10.1159/000056341. PMID 11316970
- [Background] Vierkotter A, Ranft U, Kramer U, Sugiri D, Reimann V, Krutmann J. The SCINEXA: a novel, validated score to simultaneously assess and differentiate between intrinsic and extrinsic skin ageing. J Dermatol Sci. 2009 Mar;53(3):207-11. doi: 10.1016/j.jdermsci.2008.10.001. Epub 2008 Dec 6. PMID 19059763